CLINICAL TRIAL: NCT04528082
Title: A Phase 3, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group Study, Followed by an Active Treatment Phase to Evaluate the Efficacy and Safety of Apremilast in Children From 2 to Less Than 18 Years of Age With Active Oral Ulcers Associated With Behçet's Disease (BEAN)
Brief Title: Apremilast Pediatric Study in Children With Active Oral Ulcers Associated With Behçet's Disease
Acronym: BEAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20190530; 2023-503436-40-00 (EU CTIS Number)
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Behçet Disease
Keywords: Behçet's Disease; Oral ulcers; Apremilast
MeSH Terms: conditions — Behcet Syndrome; Oral Ulcer | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: The participants will be randomized to receive apremilast or placebo in the double-blind 12 week treatment phase. Then, the participants will all receive apremilast for a further 40 weeks in the active treatment phase. The participants will then complete the 30 days safety follow-up period after the last dose of apremilast in the active treatment phase.
  Participants who complete the 52 weeks of treatment may have the opportunity to continue receiving apremilast through an open-label extension study (NCT05767047) . The participants who choose not to participate in the optional open-label, long-term study will complete the 30 days safety follow-up period after the last dose of apremilast in the active treatment phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Apremilast (Experimental): Participants will receive apremilast orally in the double-blind 12 week treatment phase. Then the participants will continue to receive apremilast in the active 40 weeks treatment phase.
  Interventions: Drug: Apremilast
- Placebo to Apremilast (Placebo Comparator): Participants will receive the matching placebo orally in the double-blind 12 week treatment phase. Then the participants will receive apremilast in the active 40 weeks treatment phase.
  Interventions: Drug: Apremilast; Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Participants will receive apremilast orally.
  Other Names: Otezla®
Drug: Placebo — Participants will receive the matching placebo orally.
  Arms: Placebo to Apremilast

SUMMARY:
The aim of this study is to estimate the efficacy of apremilast compared to placebo in the treatment of oral ulcers in pediatric participants from 2 to < 18 years of age with oral ulcers associated with Behçet's disease (BD) through week 12.

ELIGIBILITY:
Key Inclusion Criteria

* Male or Female participants 2 to < 18 years of age at randomization.
* Diagnosed with BD meeting the ISGBD criteria at any time prior to the screening visit.
* Oral ulcers that occurred ≥ 3 times within the 12-month period prior to the screening visit.
* Participant must have ≥ 2 oral ulcers at both the screening visit and on day 1.
* Participant has had prior treatment with ≥ 1 non-biologic BD therapy, such as, but not limited to, topical corticosteroids or systemic treatment.

Key Exclusion Criteria

* Behçet's disease-related active major organ involvement - pulmonary (eg, pulmonary artery aneurysm), vascular (eg, thrombophlebitis), gastrointestinal (eg, ulcers along the gastrointestinal tract), or CNS (eg, meningoencephalitis) manifestations, or ocular lesions (eg, uveitis) requiring immunosuppressive therapy; however:

  * Previous major organ involvement is allowed if it occurred ≥1 year prior to the screening visit and is not active at time of enrollment
  * Participants with mild BD-related ocular lesions not requiring systemic immunosuppressive therapy are allowed
  * Participants with BD-related arthritis and BD-skin manifestations are also allowed.
* Previous exposure to biologic therapies for the treatment of BD oral ulcers, previous biologic exposure is allowed for other indications (including other manifestations of BD).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2030-02-07 (Estimated); Study Completion 2030-12-17 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve for the Number of Oral Ulcers from Week 0 Through Week 12 (AUCw0-12) | Week 0 to Week 12

SECONDARY OUTCOMES:
Number of Oral Ulcers from Week 0 to Week 12 | Week 0 to Week 12
Change from Week 0 to Week 12 in the Pain of Oral Ulcers in Participants 5 Years of Age and Older | Week 0 to Week 12
  Pain of oral ulcers will be measured by a visual analog scale (VAS). The participants will be asked to place a vertical line on a 100 mm VAS at the point that represents the severity of oral ulcer pain. The scale will range from "no pain" (left hand boundary) to "worst possible pain" (right hand boundary).
Complete Response Rate for Oral Ulcers | Week 12
  Complete response rate for oral ulcers is defined as the proportion of participants who are oral ulcer free at Week 12.
Proportion of Participants at Week 12 Whose Number of Oral Ulcers is Reduced by Greater Than or Equal to 50% from Week 0 | Week 0 to Week 12
Complete Response Rate for Genital Ulcers | Week 12
  Complete response rate for genital ulcers is defined as the proportion of participants (with genital ulcers at week 0) who are genital ulcer free at Week 12.
Change from Week 0 to Week 12 in Disease Activity | Week 0 to Week 12
  Disease activity is measured by Behçet's Disease Current Activity (BDCAF) scores. The BDCAF consists of 3 component scores: the Behçet's Disease Current Activity Index (BDCAI) score, the Patient's Perception of Disease Activity, and the Clinician's Overall Perception of Disease Activity. The BDCAI score ranges from 0 to 12. A higher score indicates higher level of disease activity (worsening), and a negative change from baseline indicates improvement. The Patient's Perception of Disease Activity and the Clinician's Overall Perception of Disease Activity were assessed by the subject and the clinician, respectively, using a scale of 1 to 7, where a higher score indicates a higher level of disease activity.
Proportion of Participants at Week 12 Who Have New-onset or Recurrence of Behçet's-related Manifestations (Other than Oral and Genital Ulcers) | Week 12
Change from Week 0 to Week 12 on the Short Form Survey (SF-10) | Week 0 to Week 12
  The SF-10 Health Survey for Children is a parent-completed survey that contains 10 questions adapted from the Child Health Questionnaire. The SF-10 is intended to produce physical and psychosocial health summary measures. Each of the 10 questions responses is scored with a point value from 1 to 6 (1 is the worst possible condition and 6 is the best possible condition). The SF-10 physical and psychosocial measures are scored such that higher scores indicate more favorable functioning.
Number of Participants with a Treatment-emergent Adverse Event | Up to Week 56
Occurrence, Severity, and Frequency of Suicide/Suicide-related Ideations and Behaviors as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Week 56
  The C-SSRS is an assessment tool that evaluates suicidal ideation and behavior. Number of participants with suicidal ideation or behavior is defined as the number of participants who answer "yes" at any time during the study (up to end of safety follow-up, Week 56) to one of the 10 categories:
  Category 1: Wish to be dead Category 2: Non-specific active suicidal thoughts Category 3: Active suicidal ideation with any methods (not plan) without intent to act Category 4: Active suicidal ideation with some intent to act, without specific plan Category 5: Active suicidal ideation with specific plan and intent Category 6: Preparatory acts or behavior Category 7: Aborted attempt Category 8: Interrupted attempt Category 9: Actual attempt (non-fatal) Category 10: Completed suicide
Change from Week 0 to Week 52 in Tanner Staging | Week 0 to Week 52
  Tanner Staging of sexual development assessment will be used to assess sexual maturity. Tanner Staging assessment consists of 3 domains (pubic hair, breast development, and other changes) for girls and 4 domains (pubic hair, penis development, testes development, and other changes) for boys. Stages range from 1-5, with 1 indicating preadolescent and 5 adult.
Change in Body Weight Measurements | Week 0 to Week 56
Change in Height Measurements | Week 0 to Week 56
Change in Body Mass Index (BMI) | Week 0 to Week 56
  BMI assessed as weight/(height/100)^2
Plasma Concentrations of Apremilast | Up to Week 52
Taste and Acceptability of Apremilast | Week 0 and Week 2
  Taste and acceptability will be assessed using a questionnaire with a 7-point faces Likert Scale, with 1 ranging from "super bad" to 7 "super good" and questions to determine whether the participants are able to take the treatment medication.
Proportion of Participants Who Require Protocol-prohibited Medications due to Worsening of Behçet's Disease | Week 0 to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (27):
- France (3):
  - Hospices Civils de Lyon Hopital Femme Mere Enfant, Bron
  - Hopital Necker Enfants Malades, Paris
  - Hopital Robert Debre, Paris
- Greece (3):
  - Agia Sofia Children Hospital, Athens
  - Attikon University General Hospital, Athens
  - General Hospital of Thessaloniki Ippokrateio, Thessaloniki
- Meir Medical Center, Kfar Saba, Israel
- Italy (4):
  - Ospedale Santissima Annunziata, Chieti
  - IRCCS Istituto Giannina Gaslini, Genova
  - Azienda Socio Sanitaria Territoriale Centro Specialistico Ortopedico Traumatologico Gaetano Pini, Milan
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
- Spain (6):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Turkey (Türkiye) (6):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Umraniye Egitim ve Arastirma Hastanesi, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi Hastanesi, Izmir
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
- United Kingdom (3):
  - Birmingham Childrens Hospital, Birmingham
  - Alder Hey Childrens Hospital, Liverpool
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com